CLINICAL TRIAL: NCT00362050
Title: A Phase II, Double-Blind, Parallel-Group, Randomized, Dose-Ranging Study Assessing the Antimalarial Activity and Safety of RBx 11160 Administered for 7 Days in Patients With Acute Uncomplicated Plasmodium Falciparum Malaria
Brief Title: RBx11160 Phase II Dose Ranging Study RBx/MMV05-06
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medicines for Malaria Venture (Other)
Collaborators: Ranbaxy Laboratories Limited (Industry); Swiss Tropical & Public Health Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RBx/MMV05-06
Record Dates: First submitted 2006-08-08; First posted 2006-08-09 (Estimated); Last update posted 2007-08-29 (Estimated); Status verified 2007-08

CONDITIONS: Plasmodium Falciparum Malaria
Keywords: malaria, falciparum; uncomplicated Plasmodium falciparum malaria
MeSH Terms: conditions — Malaria, Falciparum | interventions — Therapeutics

INTERVENTIONS:
Drug: Treatment with 3 dose groups of RBx11160 over 7 days

SUMMARY:
The trial will identify the best dose of the synthetic peroxide RBx11160 to treat uncomplicated malaria. Patients will be treated over 7 days with daily doses of 50, 100 or 200 mg RBx11160.

The study is designed to assess the antimalarial activity and safety of 3 dose levels of RBx 11160 administered once daily for 7 consecutive days. The primary endpoint will be the time to 90% parasite clearance. In future regulatory studies, RBx 11160 is likely to be administered in combination with another antimalarial agent since the development plan follows the current recommendation of WHO for the treatment of uncomplicated malaria. However, it is critical to gather data on RBx 11160 when used as monotherapy in adult patients suffering from acute uncomplicated P. falciparum malaria. In malaria-endemic regions, an adult population is defined on the basis of immune status rather than the legal age of consent. Thus, patients as young as 13 years of age can be enrolled provided consent has been obtained from a legal guardian in accordance with local practices and regulations. This study will be conducted in compliance with International Conference on Harmonization (ICH) Good Clinical Practice (GCP).

DETAILED DESCRIPTION:
This is a Phase II, double-blind, multicenter, randomized, parallel-group, dose-ranging study of the antimalarial activity and safety of 3 (50, 100, and 200 mg) RBx 11160 dose levels administered as a single dose orally for 7 consecutive days in patients with acute uncomplicated P. falciparum malaria (mono-infection).

At least 255 patients will be randomized at 4 study sites in South East Asia, India and Africa. Each investigational site will enroll between 60 and 90 patients to yield approximately 65 "per protocol" patients in each treatment arm . Patients will be randomized to 1 of 3 dose groups. Patients will be administered RBx 11160 with matching placebo tablets as required to maintain the study blind.

The study is divided into 3 main periods including the Pre-Treatment Period (Screening/Day 0), the Treatment Period (Days 0 through 6; Day 0 is the first day of study medication dosing), and the Post-Treatment Period (Day 14 +/- 1 day; Day 21 +/- 1 day; and Day 28 +/- 2 days).

Patient participation will be for at least 28 (± 2) days following the first dose of study medication. Patients will be hospitalized for at least 4 days (Days 0, 1, 2, and 3), but may remain in the hospital or live in the vicinity of the study site for the study duration. If a patient is discharged from the hospital on Day 3, he/she will return to the study site or an authorized study staff member will visit the patient on Days 4 and 5 to administer study medication and perform indicated assessments. The patient will return to the study site for study visits on Days 6 (last dose of study medication administration), 14, 21, and 28.

If adverse events reported during the study are unresolved by Day 28, patients will be followed for an additional 30 days or until resolution of the event or determination that no further medical management is deemed necessary. Similarly, the investigator will instruct the patient to return to the study site if any untoward event occurs within 30 days of completing study medication.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 13 to 65 years, inclusive.
* Body weight > 30 kg with no clinical evidence of severe malnutrition.
* Presence of acute symptomatic uncomplicated malaria with a diagnosis confirmed by a positive blood smear with asexual forms of P. falciparum parasites only. Initial parasite densities appropriate for inclusion will be between 1000 and 100,000 asexual parasites/microL blood.
* Presence of fever (axillary temperature > 37.5 °C or oral or rectal temperature > 38 °C).
* Female patients must be non-lactating and willing to use contraceptive methods during the study period.
* Written informed consent, in accordance with local practice, provided by patient and/or parent/guardian/spouse. If a patient is unable to provide informed consent in writing, a thumbprint to indicate consent in the presence of at least 1 witness is acceptable. If applicable, for adolescents providing written informed consent, assent should be obtained from the patient's legally accepted representative/guardian.
* Willingness and ability to comply with the study protocol for the duration of the study.
* Patient resides within a reasonable distance of the investigational site, so that attendance of all study visits and follow-up by medical staff are logistically feasible.

Exclusion Criteria:

* Patients presenting with a mixed infection (i.e., malaria due to more than 1 causative parasite).
* Patients with severe malaria.
* Any antimalarial treatment during 2 weeks prior to Screening, as assessed by medical history.
* History of hypersensitivity or allergic reactions to artemisinins.
* Patients who have been treated with RBx 11160 in any study.
* Participation in any investigational drug study during the 30 days prior to Screening.
* Electrocardiogram (ECG) abnormalities with clinical significance or relevance that require urgent management. These abnormalities include QTc interval > 450 msec at Screening and cardiac conduction disorders, with the exception of right bundle branch block.
* A female patient who is lactating or pregnant at Screening.
* Gastrointestinal dysfunction that could alter absorption or motility (e.g., diarrhea defined as > 3 episodes of watery stools in the previous 24 hours or patients who have had 3 episodes of vomiting within 24 hours prior to Screening).
* Patients with known significant renal or hepatic impairment indicated by the following laboratory evaluations at Screening:

Serum creatinine > 1.5 x upper limit of normal (ULN). Aspartate transaminase > 2.5 x ULN. Alanine transaminase > 2.5 x ULN. Alkaline phosphatase > 2.5 x ULN. Total bilirubin > 1.5 x ULN.

* Patients who have had a splenectomy.
* Immunocompromised patients, patients receiving immunosuppressive agents, or patients with known human immunodeficiency virus (HIV) infection. (Screening for these conditions is not required for entry in the study.)
* Evidence of clinically significant cardiovascular, pulmonary, metabolic, gastrointestinal, neurological, psychiatric (e.g., depression, anxiety, psychosis, or schizophrenia) or endocrine diseases, malignancy, or other abnormalities (other than the indication being studied).
* Patients who have epilepsy or a history of convulsions.

Ages: 13 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 255
Dates: Start 2006-06; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Median time to 90% parasite clearance (PC90).

SECONDARY OUTCOMES:
Median time to 50% parasite clearance
Median parasite clearance time
Fever clearance time
Proportion of patients with Polymerase Chain Reaction (PCR)-corrected Adequate Clinical and Parasitological Response (ACPR) on Day 28. Proportion of patients with PCR-uncorrected ACPR on Day 28.
Proportion of patients with PCR-uncorrected ACPR on Day 14.
Relationship between RBx 11160 plasma concentrations at approximately 3 hours and 8 hours after study medication administration on Days 0 and 6 and PC90, PC50 and PCT.
Number of gametocytes at Days 0, 3, 6, 14, 21, and 28.
Safety endpoints:
Incidence of adverse events or clinically significant changes in laboratory parameters, physical examination, ECG, or vital signs.

CONTACTS AND LOCATIONS:
Overall Officials: Sornchai Looareesuwan, MD, Principal Investigator — Mahidol University; Salim M Abdulla, MD, Principal Investigator — District Hospital Bagamoyo, Dar es Salaam, Tanzania; Anders Björkman, MD, Principal Investigator — Kivunge Public Health Care Center, Zanzibar, Tanzania; Neena Valecha, MD, Principal Investigator — Malaria Research Center, Rourkela, India
Locations (4):
- Field Station Malaria Reseach Centre (Indian Council of Medical Research), Rourkela, Odisha, India
- Tanzania (2):
  - Public Health Care Center, Kivunge, Zanzibar
  - District Hospital Bagamayo, Dar es Salaam
- Faculty of Tropical Medicine, 420/6 Rajavithee Road, Bangkok, Thailand

REFERENCES:
- [Background] Vennerstrom JL, Arbe-Barnes S, Brun R, Charman SA, Chiu FC, Chollet J, Dong Y, Dorn A, Hunziker D, Matile H, McIntosh K, Padmanilayam M, Santo Tomas J, Scheurer C, Scorneaux B, Tang Y, Urwyler H, Wittlin S, Charman WN. Identification of an antimalarial synthetic trioxolane drug development candidate. Nature. 2004 Aug 19;430(7002):900-4. doi: 10.1038/nature02779. PMID 15318224
- [Background] Tang Y, Dong Y, Vennerstrom JL. Synthetic peroxides as antimalarials. Med Res Rev. 2004 Jul;24(4):425-48. doi: 10.1002/med.10066. PMID 15170591
- [Derived] Valecha N, Looareesuwan S, Martensson A, Abdulla SM, Krudsood S, Tangpukdee N, Mohanty S, Mishra SK, Tyagi PK, Sharma SK, Moehrle J, Gautam A, Roy A, Paliwal JK, Kothari M, Saha N, Dash AP, Bjorkman A. Arterolane, a new synthetic trioxolane for treatment of uncomplicated Plasmodium falciparum malaria: a phase II, multicenter, randomized, dose-finding clinical trial. Clin Infect Dis. 2010 Sep 15;51(6):684-91. doi: 10.1086/655831. PMID 20687837